CLINICAL TRIAL: NCT05386680
Title: Phase IIIb, Open-label, Single-arm, Multi-center Study to Evaluate the Safety, Tolerability and Efficacy of OAV101 Administered Intrathecally (1.2 x 10^14 Vector Genomes) to Participants 2 to < 18 Years of Age With Spinal Muscular Atrophy (SMA) Who Have Discontinued Treatment With Nusinersen (Spinraza®) or Risdiplam (Evrysdi®)
Brief Title: Phase IIIb, Open-label, Multi-center Study to Evaluate Safety, Tolerability and Efficacy of OAV101 Administered Intrathecally to Participants With SMA Who Discontinued Treatment With Nusinersen or Risdiplam
Acronym: STRENGTH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COAV101B12302
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Results first posted 2025-06-03 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Spinal Muscular Atrophy
Keywords: Zolgensma; OAV101; AVXS 101; gene therapy; Muscle atrophy; SBMA; spinal and bulbar muscular atrophy; spinal muscular atrophy; bulbar muscular atrophy; muscle function; myopathy; muscle wasting; atrophied muscle; loss of muscle strength; SMA
MeSH Terms: conditions — Muscular Atrophy, Spinal; Muscular Atrophy; Bulbo-Spinal Atrophy, X-Linked; Muscular Diseases | interventions — Zolgensma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OAV-101 (Experimental): Intrathecal administration of OAV101 at a dose of 1.2 x 10^14 vector genomes, one time dose
  Interventions: Genetic: OAV101

INTERVENTIONS:
Genetic: OAV101 — Intrathecal administration of OAV101 at a dose of 1.2 x 10^14 vector genomes, one time dose
  Other Names: AVXS-101; Zolgensma

SUMMARY:
This was a Phase IIIb open-label, single arm, multi-center study to evaluate the safety, tolerability and efficacy of OAV101B in participants with SMA aged 2 to <18 years after the discontinuation of treatment with nusinersen or risdiplam. The study aimed to enroll approximately 28 participants across each of 2 age brackets (2 to <6 years, and 6 to <18 years).

DETAILED DESCRIPTION:
Eligible participants received a single OAV101B administration of 1.2x1014 vector genomes on Day 1 (Treatment period) and were followed for a period of 52 weeks.

Participants were admitted to the hospital on Day -1 for pre-treatment baseline procedures. After receiving OAV101B on Day 1, participants underwent in-patient safety monitoring over the next 48 hours, after which the participant could be discharged, based on Investigator judgment.

ELIGIBILITY:
Inclusion Criteria

* SMA diagnosis
* Aged 2 to < 18 years
* Have had at least four loading doses of nusinersen (Spinraza®) or at least 3 months of treatment with risdiplam (Evrysdi®) at Screening
* Must have symptoms of SMA as defined in the protocol

Exclusion Criteria:

* Anti Adeno Associated Virus Serotype 9 (AAV9) antibody titer using an immunoassay is reported as elevated
* Clinically significant abnormalities in test results during screening
* Contraindications for lumbar puncture procedure
* At Baseline, participants are excluded if they received:

  * nusinersen (Spinraza®) or
  * risdiplam (Evrysdi®) within a defined timeframe
* Vaccinations 2 weeks prior to administration of OAV101
* Hospitalization for a pulmonary event, or for nutritional support within 2 months prior to Screening or inpatient major surgery planned.
* Presence of an infection or febrile illness up to 30 days prior to administration of OAV101
* Requiring invasive ventilation

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-11-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (3):
  - Boston Childrens Hospital, Boston, Massachusetts
  - Child Hosp Of The Kings Daughters, Norfolk, Virginia
  - University of Wisconsin Madison Medical School, Madison, Wisconsin
- Novartis Investigative Site, Parkville, Victoria, Australia
- Novartis Investigative Site, Leuven, Belgium
- Novartis Investigative Site, Montreal, Quebec, Canada
- France (2):
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Toulouse
- Novartis Investigative Site, Roma, RM, Italy
- Japan (2):
  - Novartis Investigative Site, Kurume, Fukuoka
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
- Novartis Investigative Site, Utrecht, Netherlands
- Novartis Investigative Site, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- [Derived] Kwon JM, Munell F, Le Goff L, Yuge K, Kato T, Cances C, De Waele L, Woodcock IR, Mercuri EM, Proud CM, Darras BT, Hayes LH, Oskoui M, Visootsak J, Williams G, Ilic A, Yang L, van der Pol WL. Intrathecal onasemnogene abeparvovec for treatment-experienced patients with spinal muscular atrophy: a phase 3b, open-label trial. Nat Med. 2025 Dec 8. doi: 10.1038/s41591-025-04119-2. Online ahead of print. PMID 41360995
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2618
- See also: A Pediatric Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/ppatientsummary/ppatientsummaries?periodicPatientSummaryId=698

RESULTS

PARTICIPANT FLOW:
Groups:
- OAV101 1.2x1014 vg - All Participants: Intrathecal administration of OAV101 at a dose of 1.2 x 10^14 vector genomes, one time dose
Period: Overall Study
Arm/Group | OAV101 1.2x1014 vg - All Participants
Started | 27
Completed | 25
Not Completed | 2
Not completed — Guardian decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | OAV101 1.2x1014 vg - All Participants
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.40 (3.348)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 1
  Unknown or Not Reported | 7

OUTCOME MEASURES:

1. Primary Outcome: Overview of Treatment-emergent Adverse Events by Age Subgroup
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a clinical investigation participant after providing written informed consent for participation in the study. The occurrence of AEs must be sought by non-directive questioning of the participant at each visit during the study. Adverse events also may be detected when they are volunteered by the participant during or between visits or through physical examination findings, laboratory test findings, or other assessments.
Time Frame: Adverse events were reported from single dose of study treatment plus 52 weeks, up to a maximum time period of 52 weeks.
Population: Full analysis set - all treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | OAV101 1.2x1014 vg - All Participants
Number analyzed (Participants) | 27
Participants
  Any treatment-emergent adverse event | 27
  Any treatment-emergent adverse event related to study treatment | 13
  Any serious treatment-emergent adverse event | 4
  Any serious treatment-emergent adverse event related to study treatment | 0
  Any severe treatment-emergent adverse event | 1
  Any treatment-emergent adverse event leading to study discontinuation | 0
  Any treatment-emergent adverse event leading to death | 0
  Any treatment-emergent adverse event of special interest | 13

2. Primary Outcome: Treatment-emergent Adverse Events Related to Treatment by System Organ Class, Preferred Term, Age Subgroup (>= 10%)
Description: as for outcome 1
Time Frame: Adverse events were reported from single dose of study treatment plus 52 weeks, up to a maximum time period of 52 weeks.
Population: Full analysis set - all treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | OAV101 1.2x1014 vg - All Participants
Number analyzed (Participants) | 27
Participants
  Number of participants with at least one event | 13
  Gastrointestinal disorders | 7
  -Vomiting | 6
  General disorders and administration site conditions | 5
  -Pyrexia | 3
  Nervous system disorders | 6
  -Headache | 4

3. Primary Outcome: Adverse Events of Special Interest by System Organ Class, Preferred Term, Age Subgroup
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a clinical investigation participant after providing written informed consent for participation in the study. The occurrence of AEs must be sought by non-directive questioning of the participant at each visit during the study. Adverse events also may be detected when they are volunteered by the participant during or between visits or through physical examination findings, laboratory test findings, or other assessments.
  An adverse event of special interest (AESI) is primarily defined by using standard Medical Dictionary for Regulatory Activities (MedDRA) queries, and identified as follows: Hepatotoxicity, Transient thrombocytopenia, Thrombotic microangiopathy, Cardiac adverse events, signs and symptoms that may be suggestive dorsal root ganglia toxicity, and new malignancies.
Time Frame: Adverse events were reported from single dose of study treatment plus 52 weeks, up to a maximum time period of 52 weeks.
Population: Full analysis set - all treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | OAV101 1.2x1014 vg - All Participants
Number analyzed (Participants) | 27
Participants
  Hepatotoxicity - Number of participants with at least one event | 4
  -Hepatic enzyme increased | 3
  -Hypertransaminasaemia | 1
  Transient thrombocytopenia - Number of participants with at least one event | 8
  -Epistaxis | 3
  -Contusion | 2
  -Bone contusion | 1
  -Gastric haemorrhage | 1
  -Lower gastrointestinal haemorrhage | 1
  -Petechiae | 1
  Signs of dorsal root ganglia toxicity - No. of pts. with at least one event | 2
  -Paraesthesia | 1
  -Sensory disturbance | 1
  Thrombotic microangiopathy - Number of participants with at least one event | 0
  Cardiac adverse events - Number of participants with at least one event | 0
  New malignancies - Number of participants with at least one event | 0

4. Secondary Outcome: Change From Baseline at Week 52 Visit in the HFMSE Total Score - Mean (SD)
Description: The Hammersmith Functional Motor Scale Expanded (HFMSE) is a SMA-specific 33-item assessment that is administered by qualified clinical evaluators. Each motor skill item is scored on a 3-point Likert scale from 0 (no response) to 2 (full response), with a total score range of 0 to 66. A higher score indicates a higher ability level.
Time Frame: Baseline, Week 52
Population: Full analysis set - for all treated participants with a valid measurement without a protocol deviation with impact
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | OAV101 1.2x1014 vg - All Participants
Number analyzed (Participants) | 21
scores on a scale | 0.17 (2.878)

5. Secondary Outcome: Change From Baseline at Week 52 Visit in the HFMSE Total Score - LS Means
Description: as for outcome 4
Time Frame: Baseline, Week 52
Population: Full analysis set - for all treated participants with a valid measurement without a protocol deviation with impact
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | OAV101 1.2x1014 vg - All Participants
Number analyzed (Participants) | 21
scores on a scale | 1.05 [-0.21 to 2.32]

6. Secondary Outcome: Change From Baseline at Week 52 Visit in the RULM Total Score - Mean (SD)
Description: The Revised Upper Limb Model (RULM) is a validated, SMA-specific assessment that measures motor performance in the upper limbs from childhood through adulthood in ambulatory and never ambulatory individuals with SMA. The revised version of the test consists of 19 scorable items: 18 items scored on a 0 (unable) to 2 (full achievement) scale, and one item that is scored from 0 (unable) to 1 (able). These item scores are summed to give a total score ranging from 0 to 37 points with lower scores reflecting poorer ability.
Time Frame: Baseline, Week 52
Population: Full analysis set - for all treated participants with a valid measurement without a protocol deviation with impact
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | OAV101 1.2x1014 vg - All Participants
Number analyzed (Participants) | 21
scores on a scale | 0.29 (2.849)

7. Secondary Outcome: Change From Baseline at Week 52 Visit in the RULM Total Score - LS Means
Description: as for outcome 6
Time Frame: Baseline, Week 52
Population: Full analysis set - for all treated participants with a valid measurement without a protocol deviation with impact
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | OAV101 1.2x1014 vg - All Participants
Number analyzed (Participants) | 21
scores on a scale | 0.59 [-0.56 to 1.73]

8. Secondary Outcome: Change From Baseline at Week 52 Visit in Assessment of Caregiver Experience in ACEND Instrument Score - Mean (SD)
Description: The Assessment of Caregiver Experience in Neuromuscular Disease (ACEND) instrument quantifies the caregiver impact experienced by parents/caregivers of children affected with severe neuromuscular diseases, including children with SMA. The total score is on a scale of 0 to 100 with a higher score indicating that caregivers experienced less intense caregiving impact.
Time Frame: Baseline, Week 52
Population: Full analysis set - for all treated participants with a valid measurement without a protocol deviation with impact
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | OAV101 1.2x1014 vg - All Participants
Number analyzed (Participants) | 24
scores on a scale | 1.43 (9.318)

9. Secondary Outcome: Change From Baseline at Week 52 Visit in Assessment of Caregiver Experience in ACEND Instrument Score - LS Means
Description: as for outcome 8
Time Frame: Baseline, Week 52
Population: Full analysis set - for all treated participants with a valid measurement without a protocol deviation with impact
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | OAV101 1.2x1014 vg - All Participants
Number analyzed (Participants) | 24
scores on a scale | 1.06 [-2.90 to 5.02]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from single dose of study treatment plus 52 weeks, up to a maximum time period of 52 weeks.
Arm/Group | OAV101 1.2x1014 vg - All Participants
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 4/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OAV101 1.2x1014 vg - All Participants (N=27)
Cyclic vomiting syndrome (Gastrointestinal disorders) | 1
Pyrexia (General disorders and administration site conditions) | 1
Bronchitis viral (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pneumonia aspiration (Infections and infestations) | 1
Influenza virus test positive (Investigations) | 1
Headache (Nervous system disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OAV101 1.2x1014 vg - All Participants (N=27)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 3
Toothache (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 13
Fatigue (General disorders and administration site conditions) | 4
Pyrexia (General disorders and administration site conditions) | 13
Swelling face (General disorders and administration site conditions) | 2
COVID-19 (Infections and infestations) | 4
Ear infection (Infections and infestations) | 4
Influenza (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 15
Upper respiratory tract infection (Infections and infestations) | 3
Contusion (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 3
Hepatic enzyme increased (Investigations) | 3
Weight increased (Investigations) | 5
Decreased appetite (Metabolism and nutrition disorders) | 2
Increased appetite (Metabolism and nutrition disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Scoliosis (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 8
Tremor (Nervous system disorders) | 4
Affect lability (Psychiatric disorders) | 3
Initial insomnia (Psychiatric disorders) | 2
Irritability (Psychiatric disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/80/NCT05386680/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-05): https://cdn.clinicaltrials.gov/large-docs/80/NCT05386680/SAP_001.pdf